CLINICAL TRIAL: NCT04394871
Title: An Observational Study to Assess Clinical Manifestations and Biomarkers in Amyotrophic Lateral Sclerosis Type 4, Other Inherited Neurological Disorders With RNA Processing Defects, and Other Neurological Diseases With a Gain of Function Mechanism.
Brief Title: Clinical Manifestations and Biomarkers in Amyotrophic Lateral Sclerosis Type 4 and Other Inherited Neurological Disorders of RNA Processing
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200064; 20-N-0064
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11-25

CONDITIONS: Amyotrophic Lateral Sclerosis Type 4; Inherited Neurological Disorders of RNA Processing
Keywords: Natural History Study; Biomarker Development; Natural History
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis 4, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ALS4 Patients: Patients with ALS4 inherited defect in the senataxin (SETX) gene.
- Disease Control Participants: Disease control participants with mutation in other genes which alter RNA processing (e.g., RNASEH1+2 and loss of function SETX mutations in patients with ataxia and oculomotor apraxia type 2[AOA2]).
- Gain of Function: patients with gain of function mutations in genes that result in other forms of neurological disease, as well as select patients with mutation in the SETX gene (select ALS4 patients), will be enrolled and followed annuallt for 5 years.
- Related, Unaffected Healthy Controls: Unrelated, unaffected healthy relatives of the ALS4 and disease control groups enrolled as controls.
- Unrelated, Healthy Controls: Unrelated, healthy volunteers who are age and sex matched to the affected ALS4 and disease control participants.

SUMMARY:
Background:

Amyotrophic lateral sclerosis type 4 (ALS4) is an inherited motor neuron disease. People with ALS4 have a change in the amount of RNA and DNA that bind together. This binding of RNA with DNA forms units called R-loops. Researchers want to learn how R-loops are related to ALS4. To do this, they will study people with inherited neurological conditions that may affect R-loop levels. These include ALS4, progressive external opthalmoplegia with mitochondrial deletions (PEOB2), Aicardi-Goutieres syndrome (AGS), and ataxia and oculomotor apraxia type 2 (AOA2).

Objective:

To learn how the binding of RNA with DNA (R-loops) is related to neurological disease.

Eligibility:

People age 5 and older with ALS4, PEOB2, AGS, and AOA2. Healthy relatives and nonrelatives are also needed.

Design:

Participants may be screened with a review of x-rays and other medical records.

Healthy relative and nonrelative participants will have 1 visit. All other participants will have 4 visits over 3 years.

At visits, participants will undergo some or all of the following:

Medical history

Physical exam

Tests of muscle strength and volume and physical function

Blood tests

Pregnancy test (for some females)

Skin biopsy of forearm

Magnetic resonance imaging (MRI)

Dual x-ray absorptiometry (DEXA).

Some tests are optional.

The MRI uses a magnetic field and radio waves to take pictures. Participants will lie on a table that slides in and out of the scanner. The scanner makes noise. They will get earplugs.

The DEXA scan uses x-rays to take pictures.

MRI and DEXA will be used to measure muscle, fat, and lean body mass.

...

DETAILED DESCRIPTION:
Objective:

Amyotrophic lateral sclerosis type 4 (ALS4) is an inherited form of motor neuron disease caused by a gain of function mutation in the senataxin (SETX) gene. The main goal of this study will be to collect clinical and molecular biomarkers from patients with ALS4 and other neurological diseases that have a gain of function mechanism to understand the natural history and progression of these diseases. The biomarkers identified will serve as potential tools for the evaluation of efficacy in future therapeutic studies in ALS4 and other neurological diseases that have a gain of function mechanism.

For the Inherited Forms of RNA Metabolism cohort, patients with mutation in the SETX gene (ALS4 RNA Metabolism patients) will be enrolled and followed annually for 3 years. Individuals with mutation in genes that are predicted to result in a similar disruption of RNA processing (such as ribonuclease H1 and H2 (RNASEH1+2) genes and recessive mutations in SETX will serve as disease controls and participate in follow-up for 3 years to collect clinical and molecular biomarkers. ALS4 and disease control subjects who have had their mutation identified in protocol 00-N-0043 or protocol 12-N-0095, or those who have had previous genetic testing will be potential candidates for enrollment in this study. Healthy control populations (related, unaffected healthy controls and unrelated, healthy controls) will be screened for under this study and participate in a single visit to collect clinical and molecular biomarkers. Healthy control populations will participate in clinical and molecular biomarker collection for comparison to all ALS4 patients in study. Related, unaffected healthy controls may also be screened under protocol 00-N-0043. No clinical genetic testing will take place under this protocol; however, research testing of genetic modifiers may be performed.

For the Gain of Function cohort, patients with gain of function mutations in genes that result in other forms of neurological disease, as well as select patients with mutation in the SETX gene (select ALS4 patients), will be enrolled and followed annually for 5 years. Subjects in the Gain of Function cohort who have had their mutation identified in protocol 00-N-0043 or protocol 12-N- 0095, or those who have had previous genetic testing will be potential candidates for enrollment in this study. No clinical genetic testing, such as whole genome or whole exome sequencing, will take place under this protocol; however, research testing of genetic modifiers may be performed. An additional goal of this study is to share clinical and molecular measures which are sensitive at detecting disease progression with collaborators working to develop therapeutics in patients with other forms of neurological disease caused by gain of function mechanisms.

Study population:

There will be a total of 330 subjects enrolled under this protocol.

For the Inherited Forms of RNA Metabolism cohort, up to 65 participants with mutation in SETX (ALS4 RNA Metabolism patients) will be enrolled for annual follow-up, and up to 50 disease control participants with mutation in other genes which alter RNA processing (e.g., RNASEH1+2 and loss of function SETX mutations in patients with ataxia and oculomotor apraxia type 2[AOA2]) will be enrolled. Up to 150 related, unaffected healthy relatives of the ALS4 RNA Metabolism patients and disease control group may also be enrolled as controls. Additionally, a maximum of 50 unrelated healthy volunteers who are age and sex matched to the affected ALS4 RNA Metabolism patients and disease control participants will also be enrolled.

For the Gain of Function cohort, up to 15 patients with gain of function mutations in genes that result in neurological disease (including select ALS4 patients) will be enrolled.

Study Design:

For the Inherited Forms of RNA Metabolism cohort, patients with ALS4 inherited defect in SETX (ALS4 RNA Metabolism patients) will be evaluated at the NIH clinical center to characterize clinical features of the disease and collect clinical and molecular biomarkers. Disease controls will be evaluated to collect molecular biomarkers and clinical measurements at the discretion of the investigator. ALS4 RNA Metabolism patients and Disease Control participants will report to the NIH every 12 months ( 60 days) for clinical and molecular studies for a total of 4 visits. Healthy control populations (related, unaffected healthy controls and unrelated healthy controls) will be evaluated for a single visit to collect clinical and molecular biomarkers. An offsite visit, conducted in person at the participant s home, may be completed for the related, unaffected healthy control group, the disease control group, and in up to 15 ALS4 RNA Metabolism participants in the Inherited Forms of RNA Metabolism cohort.

For the Gain of Function cohort, patients with gain of function mutations and neurological disease (including select SETX/ALS4 patients) will be evaluated at the NIH clinical center for a time period up to 5 years at a frequency determined by the discretion of the investigator, but no more frequent than every 6 months, for a total of up to 11 visits. Participants in the Gain of Function cohort will not be seen offsite.

Outcome measures:

No specific primary and secondary outcomes will be specified; however, the change in the following measures from baseline may be used to characterize the baseline status and disease progression and disease severity over the course of the study.

For both the Inherited Forms of RNA Metabolism cohort and the Gain of Function cohort: neuromuscular ultrasound, magnetic resonance imaging (MRI) evaluation of the lower extremity (muscle volume and fat fraction), dual-energy X-ray absorptiometry (DEXA) scan of whole body composition (lean body mass), quantitative muscle strength testing (QMT) of the upper and lower extremities, 6 minute timed walk test (6MTWT), timed up and go (TUG), 30 second chair stand test, pinch strength test, activity card sort (ACS), disabilities of the arm, shoulder, and hand (DASH), SF36 questionnaire, ALS Health Index (ALS-HI) questionnaire, Patient-Perceived Change in Function Question, Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSAQ-5), and the grooved pegboard test.

Molecular biomarkers will be evaluated in ALS4 patients (from both the Inherited Forms of RNA metabolism cohort and the Gain of Function cohort) and in the control groups (healthy and disease) (from the Inherited Forms of RNA metabolism cohort) to identify those molecular biomarkers that are disease specific (disease vs. control) as well as those that are informative of disease progression in ALS4 (early vs. advanced disease).

For the Gain of Function cohort, the following additional measures may be used: revised upper limb module (RULM); Myotools assessment; 32 item motor function measure (MFM32); 9-hole peg test; Charcot-Marie-Tooth functional outcome measure (CMT-FOS); nerve conduction studies; electrical impedence myography (EIM); and accelerometry assessment.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALS4 RNA metabolism inclusion criteria:

* Age 5 or above
* Genetic diagnosis of ALS4 (heterozygous mutation in SETX)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Capacity to consent (adults) or assent (pediatric subjects) to the study

Disease control inclusion criteria:

* Age 5 or above
* Genetic diagnosis of RNA processing defect mutation (RNaseH1, RNaseH2, recessive mutations in SETX)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Capacity to consent (adults) or assent (pediatric subjects) to the study

Related, unaffected healthy control inclusion criteria:

* Age 5 or above
* Family history (first, second, or third degree relative) of RNA processing defect mutation (RNaseH1, RNaseH2, heterozygous or recessive mutations in SETX)
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Capacity to consent (adults) or assent (pediatric subjects) to the study

Unrelated, healthy control inclusion criteria:

* Age 5 or above
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Capacity to consent (adults) or assent (pediatric subjects) to the study

Gain of function inclusion criteria:

* Age 5 or above
* Genetic diagnosis of mutation resulting in a gain of function mechanism (for example, heterozygous mutations in SETX or heterozygous mutations in KCC3)
* Able to communicate well with the investigator, to understand and comply with the requirements of the studyCapacity to consent (adults) or assent (pediatric subjects) to the study
* Capacity to consent (adults) or assent (pediatric subjects) to the study

EXCLUSION CRITERIA:

ALS4 RNA metabolism exclusion criteria:

* Patients with known claustrophobia, presence of pacemaker, ferromagnetic material in their body, or any other condition that would preclude MRI assessments
* Pregnancy

Note: An Adult RNA metabolism ALS4 Patient who meets any of the following criteria will be excluded from the lumbar puncture procedure:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

  * Disease control exclusion criteria:

    --Pregnancy
  * Related, unaffected healthy control exclusion criteria:

    * Diagnosis of neuromuscular disease or weakness on physical examination
    * Pregnancy

Note: An Adult Related, Unaffected Healthy Control who meets any of the following criteria will be excluded from the lumbar puncture procedure:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

  * Unrelated, healthy control exclusion criteria:

    * Diagnosis of neuromuscular disease or weakness on physical examination
    * Patients with known claustrophobia, presence of pacemaker, ferromagnetic material in their body, or any other condition that would preclude MRI assessments
  * Pregnancy

Note: An Adult Unrelated, Healthy Control who meets any of the following criteria will be excluded from the lumbar puncture procedure:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

Gain of function exclusion criteria:

-Pregnancy

Note: An Adult Gain of Function patient who meets any of the following criteria will be excluded from the lumbar puncture procedure:

* PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of normal (including treatment with oral and parenteral anticoagulants)
* INR greater than or equal to 1.5, thrombocytopenia (<70,000), or abnormal bleeding time or platelet dysfunction
* History of a bleeding disorder
* Use of anticoagulants

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Disease cohorts with defined mutations
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2030-12-25 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression as measured by thigh muscle volume and other study measures | Baseline and annually at visits 2 - 4
  Clinical and molecular measurements in ALS4 patients and other inherited neurological disorders of RNA processing will be assessed over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grunseich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rabin BA, Griffin JW, Crain BJ, Scavina M, Chance PF, Cornblath DR. Autosomal dominant juvenile amyotrophic lateral sclerosis. Brain. 1999 Aug;122 ( Pt 8):1539-50. doi: 10.1093/brain/122.8.1539. PMID 10430837
- [Background] Grunseich C, Wang IX, Watts JA, Burdick JT, Guber RD, Zhu Z, Bruzel A, Lanman T, Chen K, Schindler AB, Edwards N, Ray-Chaudhury A, Yao J, Lehky T, Piszczek G, Crain B, Fischbeck KH, Cheung VG. Senataxin Mutation Reveals How R-Loops Promote Transcription by Blocking DNA Methylation at Gene Promoters. Mol Cell. 2018 Feb 1;69(3):426-437.e7. doi: 10.1016/j.molcel.2017.12.030. Epub 2018 Jan 27. PMID 29395064
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-N-0064.html